CLINICAL TRIAL: NCT06741605
Title: Biomechanical Risk Factors of Cervical Pain in Pregnant Women
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Ahmed Ibrahim Fadel, Principal investigator, Cairo University
Other Study IDs: P.T.REC/012/005381
Record Dates: First submitted 2024-12-15; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Cervical Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women with cervical pain: Pregnant women with cervical pain in their third trimester will be assessed to investigate the relationship between biomechanical risk factors and neck pain in pregnant women.

INTERVENTIONS:
Other:

SUMMARY:
The purpose of the study is to assess the biomechanical risk factors for neck pain in pregnant women.

DETAILED DESCRIPTION:
Neck pain during pregnancy has significant physical, psychological, and social impacts on women's lives. Moreover, the economic burden of neck pain is remarkable and includes treatment costs, reduced productivity, and job-related problems. Untreated neck pain during pregnancy can potentially lead to chronic musculoskeletal problems postpartum.

The significance of the study is based on the concept of "early prediction for early mitigation of the risk and prevention of the onset or progression".

Studies have investigated risk factors for neck pain. However, there is a notable gap in research regarding these factors in pregnant women, especially physical (biomechanical) risk factors, despite the significant biomechanical changes they undergo during pregnancy. This study aims to fill this gap by investigating the relationship between biomechanical risk factors and neck pain in pregnant women.

To our knowledge, this is the first study in which this relationship will be assessed to provide evidence about the biomechanical risk factors for neck pain in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in their third trimester suffering from cervical pain.
* They have experienced cervical pain starting during pregnancy.
* They reported no neck pain or neck-related disorders during the previous year and were screened for the absence of cervical pathology during a physical examination.

Exclusion Criteria:

* Objective signs of structural pathology on physical examination, including but not limited to shoulder bursitis, impingement, tendonitis, fracture, cervical nerve or disc impairment, radiculopathy, or loss of upper extremity sensory or motor function.
* Acute injury of the neck or shoulders (<12 weeks before the study).
* History of fibromyalgia or musculoskeletal pain present in more than 4 body regions concurrently.
* Self-reported systemic illness, including cancer, rheumatic, cardiovascular, or neurological disease
* Untreated psychiatric condition
* Previous surgery involving the cervical spine or shoulders
* Uncontrolled hypertension (resting systolic blood pressure >150 mm Hg, or diastolic blood pressure >90 mm Hg).

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: They will be selected from the departments of obstetrics and gynecology at Sinhout Hospital and Minya Elkamh Central Hospital, El-Sharqia Governorate, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-02-20 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 2 months
  The VAS will be used to assess cervical pain for each pregnant woman. It is a pain rating scale, whose scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and "worst pain" on the right end of the scale (10 cm).
Measurement of trigger points | 2 months
  Pressure algometer will be used to assess the trigger points of the neck muscles of each pregnant woman in the study.
  It will be placed perpendicularly to the fibers of the upper trapezius muscle, bilaterally, exactly over the myofascial trigger points. These points were pressed until the pain is reported, and the value displayed on the equipment's display will be recorded in kg/cm2.

SECONDARY OUTCOMES:
Measurement of craniovertebral angle (CVA) | 2 months
  Posture screen analysis mobile application will be used to measure the CVA for each pregnant woman The CVA is the best indicator of forward head posture. To determine this angle, two references are defined: One line runs from the swallow of the ear to the seventh cervical vertebra (C7) and another horizontal line parallel to the ground passes only through the spinous apophysis of C7. An angle of less than 50°-53° may indicate FHP. Thereby, the smaller the CVA, the greater the disability
Measurement of cervical flexion range of motion (ROM) | 2 months
  Place the goniometer's axis over the external auditory meatus before using it. Place the stationary arm perpendicular to the floor or vertically. Place the movable arm in line with the nose's base. This should be noted as 0°.
  To assess cervical flexion: ask the patient to nod forward and bring their chin towards their chest. Normal cervical flexion is usually approximately 80º
Measurement of cervical extension range of motion (ROM) | 2 months
  Place the goniometer's axis over the external auditory meatus before using it. Place the stationary arm perpendicular to the floor or vertically. Place the movable arm in line with the nose's base. This should be noted as 0°.To assess cervical extension: ask the patient to look upwards as far as possible, until full extension of the neck is achieved. Normal cervical extension is usually 50°.
Measurement of cervical lateral flexion range of motion (ROM) | 2 months
  The goniometer fulcrum will be aligned over the spinous process of the C7. The fixed arm of the goniometer will be aligned vertically along the imaginary line between the two acromion processes. The movable arm will be aligned over the external occipital protuberance.
  Ask the patient to tilt his/her head laterally to the left, without rotating the head, while her shoulders remain fix. Repeat the procedure for the opposite side and note the angle of flexion of the head. Normal flexion from starting point on either side is 45°
Measurement of cervical rotation range of motion (ROM) | 2 months
  The goniometer fulcrum will be aligned over the center of the subject's head, the fixed arm of the goniometer will be aligned with an imaginary line between the subject's acromion processes and the movable arm will be aligned with the tip of the subject's nose.
  Ask the patient to rotate his/her head to the left as far as possible without tilting or tipping his/her head. Stabilize the shoulders by lightly pressing onto them. Repeat the process for the opposite direction. Normal rotation is approximately 80°.
Assessment of neck disability | 2 months
  The neck disability index will be used to assess neck disability for each pregnant woman. It is a well-validated 10-item questionnaire, with each item rated on a 0 to 5-point scale. The sum of the 10 items gives a score between 0-50. The lower the score, the less self-rated the disability. 0-4 = no disability, 5-14 = mild disability, 15-24 = moderate disability, 25-34 = severe disability, and 35 or over = complete disability
Measuring breast size | 2 months
  The breast size will be measured by using tape around torso on the level of the nipple to determine if breast size is a risk factor for cervical pain.

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Hussien, Professor, Study Director — Al-Azhar University; Doaa Osman, Professor, Study Chair — Cairo University
Locations (1):
- Doaa Ahmed Fadel, Zagazig, Egypt